CLINICAL TRIAL: NCT04266535
Title: TCI vs Manually Controlled Infusion of Propofol in Patients Sceduled for Laparoscopic Surgery; a Case-control Study
Brief Title: TCI vs Manually Controlled Infusion of Propofol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Regional Hospital West Jutland (Other)
Responsible Party: Principal Investigator, Niels Peter Ekeløf, Principal Investigator, Regional Hospital West Jutland
Other Study IDs: TCI/RHWJ
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia, Intravenous; Laparotomy; Airway Extubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- TCI: Patients receiving Target Controlled Infusion (TCI) Anesthesia
  Interventions: Device: Target controlled infusion
- MCI: Patients receiving Manually Controlled Infusion (MCI) Anesthesia
  Interventions: Device: Target controlled infusion

INTERVENTIONS:
Device: Target controlled infusion — Target controlled infusion vs manually controlled infusion

SUMMARY:
Anesthesia records for patients anesthetized with target controlled infusion of propofol and remifentanil will be matched with patients anesthezied with manyally controlled infusion.

The aim of the study is to verify differences in time to extubation and amount of drugs used.

anesthetize

ELIGIBILITY:
Inclusion Criteria:

- Patients to laparoscopic surgery

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anestectic records
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Post procedural awakening | 10 minutes
  Time from the surgical procedure has ended until arrival at the post anesthesia unit (PACU)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR